CLINICAL TRIAL: NCT06088836
Title: Impact of Ultrasound- Guided Continuous Retro Laminar Block Versus Continuous Erector Spinae Plane Block on Incentive Spirometry Volumes and Pain Scores in Multiple Rib Fractures
Brief Title: Ultrasound- Guided Continuous Retro Laminar Block Versus Continuous Erector Spinae Plane Block in Multiple Rib Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hossam Ibrahim Elsayed Ibrahim, Assistant Lecturer of Anesthesia, Surgical ICU and Pain Medicine Master's degree of Anesthesia, Surgical ICU And Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MD35/2/23
Record Dates: First submitted 2023-10-03; First posted 2023-10-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Retrolaminar Block; Erector Spinae Plane Block; Spirometry; Pain; Multiple Rib Fractures
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Retrolaminar block group) (Experimental): Patients received ultrasound guided Retrolaminar block bolus dose of 20 ml 0.25% bupivacaine then continuous infusion at a rate of 0.1 mL/kg/hr. for 4 days
  Interventions: Drug: Retrolaminar block group
- Group II (Erector spinae plane block group) (Experimental): Patients received ultrasound guided Erector spinae plane block bolus dose of 20 ml 0.25% bupivacaine then continuous infusion at a rate of 0.1 mL/kg/hr. for 4 days
  Interventions: Drug: Erector spinae plane block group.

INTERVENTIONS:
Drug: Retrolaminar block group — Under complete aseptic precautions and sterilization and in sitting position, A high-frequency linear ultrasound probe (6-11 MHz) was placed into a longitudinal orientation in the paraspinous line 1 cm from the midline. Lamina appeared as a continuous line interrupted by the intra laminar spaces.
  local infiltration of needle insertion site with 3ml of 2.0 % lidocaine was done Then, an 18-gauge Tuohy needle was inserted in plane 1 cm lateral to the spinous process using ultrasound imaging and advanced caudally or cranially until it contacts the lamina.
  Arms: Group I (Retrolaminar block group)
Drug: Erector spinae plane block group. — Under complete aseptic precautions and sterilization and in sitting position, A high-frequency ultrasound transducer was placed in a longitudinal orientation 3 cm lateral to the midline midway between the uppermost and the lowest fractured rib to identify counting of ribs using ultrasound three muscles were identified as superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. However, when the rhomboid major muscle disappears this indicates that we are at the level of the seventh thoracic vertebra.
  local infiltration of needle insertion site with 3ml of 2.0 % lidocaine was done. Then, an 18-gauge Tuohy needle was inserted in cranial-caudal direction towards transverse process (TP) in-plane to the US transducer until needle touched the TP crossing all the muscles
  Arms: Group II (Erector spinae plane block group)

SUMMARY:
The aim of this study is to compare the incentive spirometry volume and analgesic efficacy of ultrasound guided continuous Retrolaminar block and continuous Erector spinae plain block in patients with multiple rib fractures.

DETAILED DESCRIPTION:
Thoracic epidural analgesia (TEA) and thoracic paravertebral block (TPVB) are strongly recommended techniques for managing thoracic neuropathic pain However, they can be technically challenging to perform and are associated with up to 15% failure rate in Thoracic epidural analgesia (TEA)and potential risk of pneumothorax in thoracic paravertebral block (TPVB).Newer approaches have been the focus of many studies in recent years; these approaches include retrolaminar block and erector spinae plane block.

Retrolaminar block (RLB) is a new thoracic truncal block for controlling somatic pain in both the thoracic and abdominal walls.

The Erector Spinae plane block (ESPB) has been used successfully to manage severe neuropathic pain arising from ribs .The basis to use ESPB is its likely site of action which is the dorsal and ventral rami of the thoracic spinal nerves.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old.
* Both sexes.
* Patients with unilateral multiple traumatic rib fractures (≥ 3 ribs).

Exclusion Criteria:

* 1st ken refusal.
* Patients with any contraindication for regional block as:

  * Bleeding disorders.
  * Infection at the injection site.
  * Patients with hemodynamic instability.
* Patients with known hypersensitivity to the study drugs
* Unconscious patients
* Patients with significant trauma outside the chest wall e.g., acute spine or pelvic fracture, severe traumatic brain or spinal cord injury, or abdominal visceral injuries
* Patients with significant lung contusions, pneumothorax, flail chest
* Chronic opioid users.
* Uncooperative patients and patients with psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Maximum inspired volume | 4 days after intervention.
  Maximum inspired volume will be measure by incentive spirometry which indicate less pain.
  Inspiratory capacity (IC) measured by Incentive Spirometry before the block, 30 minutes, 60 minutes after the blocks and then every six hours for subsequent 4 days.

SECONDARY OUTCOMES:
Daily and total rescue analgesics consumption. | 24 hours after intervention.
  Need for rescue analgesia and the total consumption of morphine in the form of incremental doses (0.05mg /kg) if Visual Analogue Score (VAS) ≥4 Pain score will be measured by Visual Analogue Score (VAS) from 0 to 10. Where 0: no pain, 10: the worst pain
Intensive care length of stay. | 28 days after intervention
  Time from admission till Intensive care discharge
Hospital length of stay. | 28 days after intervention
  Time from admission till Hospital discharge
pH | 4 days after intervention.
  pH will be measure before the block ,6 hours after the block and then daily for subsequent 4 days.
PaO2 | 4 days after intervention.
  PaO2 will be measure before the block ,6 hours after the block and then daily for subsequent 4 days.
PaCo2 | 4 days after intervention.
  PaCo2 will be measure before the block ,6 hours after the block and then daily for subsequent 4 days.
FiO2 | 4 days after intervention.
  FiO2 will be measure before the block ,6 hours after the block and then daily for subsequent 4 days.
Respiratory rate | 4 days after intervention.
  Respiratory rate will be measure before the block ,6 hours after the block and then daily for subsequent 4 days.
Adverse effects and complications. | 4 days after intervention.
  Adverse effects and complications such as hypotension, complications related to catheter insertion, pneumothorax, local anesthetic toxicity, and respiratory depression

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.